CLINICAL TRIAL: NCT03264053
Title: Socket Shield Technique Versus Conventional Immediate Implant Placement in Thin Buccofacial Bone to Evaluate Buccal Bone Resorption: A Randomized Controlled Trial
Brief Title: Socket Shield Technique Versus Conventional Immediate Implant Placement in Thin Buccofacial Bone
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdullah Abdou Mattar, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-CU-2017-08-03
Record Dates: First submitted 2017-08-16; First posted 2017-08-28 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Crestal Bone Loss
Keywords: socket shield technique; crestal bone loss; immediate implanation
MeSH Terms: interventions — Immediate Dental Implant Loading

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SOCKET SHIELD TECHNIQUE (Experimental): Socket shield is the surgical removal of the frontal aspect of the badly broken root and retaining the lingual aspect so as to prevent crestal bone loss with insertion of the dental implant behind it
  Interventions: Device: Socket shield
- Conventional immediate implantation (Active Comparator): Conventional immediate implantation is the surgical removal of the entire badly broken root
  Interventions: Procedure: Conventional immediate implantation

INTERVENTIONS:
Device: Socket shield — Socket shield is the Removal of the lingual portion of the anterior root thus retaining the lingual portion
  Other Names: Implant stability
  Arms: SOCKET SHIELD TECHNIQUE
Procedure: Conventional immediate implantation — Conventional immediate implantation
  Arms: Conventional immediate implantation

SUMMARY:
Buccal bone is prone to resorb after tooth extraction specially with immediate tooth implantation which could compromise the esthetics of the patient. socket shield technique retains the buccal aspect of the extracted root fragment which may help in preventing the buccal bone from resorbing and prevent esthetics deterioration

DETAILED DESCRIPTION:
The alveolar ridge resorbs and collapses following tooth removal which continues to be a major concern for practitioners. Many researchers concluded that buccal aspect of the ridge is more prone to resorption, as it is primarily supplied by the periodontal tissues and ligments of the tooth. Therefore, extraction of the hopeless tooth, may be a reason for buccal cortical plate resorbing at a faster rate than the palatal plate leading to its total degradation. This may lead to dimensional changes in the human ridge and the aesthetic area is highly affected by this process. Several techniques in the litreture were proposed to solve the problem of thin buccal bone resorption with or without immediate implantation in the aesthetic area. Some of these techniques are the guided bone and soft tissue regenraton and bone augmentation but proved to be slight aggressive with high morbidity rate. Recently, several papers were published concerning the socket shield technique explaining how to maintain the ridge width and height. Socket shield technique that was first introduced in 2010 aids at retaining the buccal fragment of root in place and intact thus placing the implant behind the lingual aspect of that fragment so that the periodontal ligments and tissues preserve its vitality and aids in preventing the collapsing of the buccal bone. This would help in improving aesthetics especially during immediate implant placment in the anterior maxillary region.

ELIGIBILITY:
Inclusion Criteria:

* • Humans

  * Esthetic area (anterior and first premolars)
  * Intact labial plate
  * Hopeless tooth indicated for extraction and immediate implant placement

Exclusion Criteria:

* • Implantation after trauma

  * Peri-implantits defects
  * Use of barrier membranes(GBR)
  * Socket preservation

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Estimated)
Dates: Start 2017-08-20 (Actual); Primary Completion 2018-08-20 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
Buccal bone resorption assesed by cone beam computed tomography as a measuring tool | 12 months
  Measuring buccal bone loss after the procedure comparing between leaving the buccal portion of the root and extracting the whole root

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah A Mattar, A.Lecturer, Principal Investigator — Cairo University
Locations (1):
- Cairo university, Cairo, Egypt